CLINICAL TRIAL: NCT03483948
Title: A Phase I Study of Safety, Pharmacokinetics and Efficacy of HMPL-523 With Azacitidine in Elderly Patients With Previously Untreated Acute Myeloid Leukemia
Brief Title: Phase I Study of HMPL-523+Azacitidine in Elderly Patients With Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow Enrollment
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-523-00CH3
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HMPL-523 & Azacitidine (Experimental): HMPL-523 will be taken orally once daily continuously through a 28-days Cycle of study treatment. Azacitidine will be administered subcutaneously, beginning on Day 1 through Day 7 of each Cycle.
  Interventions: Drug: HMPL-523; Drug: Azacitidine

INTERVENTIONS:
Drug: HMPL-523 — HMPL-523 tablet
Drug: Azacitidine — Azacitidine Injection
  Other Names: Vidaza

SUMMARY:
This is a Phase I, open-label, non-randomized, multicenter study to evaluate the safety, pharmacokinetics and preliminary efficacy of HMPL-523 in combination with Azacitidine in previously untreated elderly patients with AML who are not eligible for standard induction therapy.

DETAILED DESCRIPTION:
There are two stages in this study: a dose-escalation stage (stage 1) and a dose-expansion stage (stage 2).

Dose-escalation stage (stage 1):

The conventional 3+3 design (3 patients per dose cohort, with the potential to add additional 3 patients to the same cohort to further evaluate toxicity) will be applied for dose escalation and maximum tolerated dosage determination. Approximately 12 to 18 dose limited toxicities evaluable patients will be enrolled. A dose of HMPL-523 up to 800mg will be taken orally once daily continuously through a 28-day Cycle of study treatment. Azacitidine will be administered subcutaneously, beginning on Day 1 through Day 7 of each Cycle.

Dose-expansion stage (stage 2):

This phase is to further evaluate the safety, pharmacokinetics and preliminary efficacy of HMPL-523 in combination with Azacitidine in approximately 28 previously untreated elderly patients with AML. Patients will receive HMPL-523 in combination with Azacitidine in a 28-day cycle continuously until disease progression/relapse, death, or intolerable toxicity, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have confirmation of AML by WHO criteria, except for APL (M3)
2. Subject must be ≥ 65 years of old and be ineligible for treatment with a standard cytarabine and anthracycline induction regimen due to co-morbidity or other factors
3. Subject must have received no prior treatment for AML with the exception of hydroxyurea
4. ECOG performance status of 0-1. For dose-expansion stage, ECOG PS of 2 will also be eligible

Exclusion Criteria:

1. Subject has received treatment of hypomethylating agent and/or chemo therapeutic agent for MDS or MPN
2. Subject has known active CNS involvement or extramedullary sarcoma from AML
3. Subject has favorable risk cytogenetics as categorized by the NCCN Guidelines Version 1, 2018 for Acute Myeloid Leukemia, such as inv(16) or t(16;16) or t(8;21) or t(15;17)
4. Subject has a white blood cell count > 25 × 109/L (Hydroxyurea is permitted to meet this criterion)
5. Subject with serum amylase or lipase > the ULN
6. Subject is known to be positive for hepatitis B or C infection with the exception of those with an undetectable viral load.
7. Subject who don't have enough liver or renal function
8. Subject with New York Heart Association (NYHA) Class III or greater congestive heart failure
9. Subject received herbal therapy ≤ 1 week prior to initiation of study treatment
10. Subject received prior treatment with any SYK inhibitors (Fostamatinib) or FLT3 inhibitor (Quizartinib) or multi-target inhibitor with SYK or FLT3 inhibition activity (Midostaurin)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Adverse Event (AE) monitoring of HMPL-523 in combination with azacitidine | Measured from the first dose to within 30 days after the last dose.
  AE monitoring will be assessed by evaluation of study drug exposure, AEs , serious AEs, all deaths, as well as laboratory determinations and vital sign parameters.
Overall response rate (ORR) | Measured up to 1 year after the last subject has enrolled or all the subjects have finished their last EFS follow up, whichever comes first.
  Overall response rate will be defined as the proportion of subjects who achieve a complete remission (CR), complete remission incomplete (CRi), Morphologic leukemia-free state (MLFS), or partial remission(PR) per 2017 European Leukemia Net (ELN) recommendations

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of HMPL-523 | Measured on the cycle 1 day 7, cycle 1 day 8, cycle 1 day 28 and cycle 2 day 1.
  Maximum concentration, occurring at Tmax.
The time to Cmax (peak time, Tmax) of HMPL-523 | Measured on the cycle 1 day 7, cycle 1 day 8, cycle 1 day 28 and cycle 2 day 1.
  The time at which maximum plasma concentration (Cmax) is observed.
The area under the plasma concentration-time curve (AUC) from 0 to the time of the last measurable concentration (AUCt) of HMPL-523 | Measured on the cycle 1 day 7, cycle 1 day 8, cycle 1 day 28 and cycle 2 day 1.
  The area under the plasma concentration-time curve (AUC) from 0 to the time of the last measurable concentration.
Half-life (t1/2) of HMPL-523 | Measured on the cycle 1 day 7, cycle 1 day 8, cycle 1 day 28 and cycle 2 day 1.
  The time required for the concentration of the drug to reach half of its original value.
Clearance (CL) of Azacitidine | Measured on the cycle 1 day 7 and Cycle 1 day 8.
  Clearance is defined as the rate at which drug is cleared from the blood.
The area under the plasma concentration-time curve (AUC) from 0 to the time of the last measurable concentration (AUCt) of Azacitidine | Measured on the cycle 1 day 7 and Cycle 1 day 8.
  The area under the plasma concentration-time curve (AUC) from 0 to the time of the last measurable concentration.
Half-life (t1/2) of Azacitidine | Measured on the cycle 1 day 7 and Cycle 1 day 8.
  The time required for the concentration of the drug to reach half of its original value.
Steady-state concentration(Css) of Azacitidine | Measured on the cycle 1 day 7 and Cycle 1 day 8.
  The average concentration of drug at steady state
Complete Remission Rate of Minimal Residual Disease (MRD) Negativity （CR MRD- rate） | Measured up to 1 year after the last subject has enrolled or all the subjects have finished their last EFS follow up, whichever comes first.
  CR MRD- rate will be defined as the proportion of subjects who achieve a CR and has a negative RT-qPCR or MFC at the same time.
Event Free Survival (EFS) | Measured up to 1 year after the last subject has enrolled or all the subjects have finished their last EFS follow up, whichever comes first.
  EFS will be defined as the number of days from the date of first dose to the date of earliest recurrence or PD or death.
Disease-free Survival (DFS) | Measured up to 1 year after the last subject has enrolled or all the subjects have finished their last EFS follow up, whichever comes first.
  DFS will be defined as the number of days from the date of composite complete response (CR + CRi) to the date of earliest recurrence or death.
Overall Survival (OS) | Measured up to 1 year after the last subject has enrolled or all the subjects have finished their last EFS follow up, whichever comes first.
  OS will be defined as the number of days from the date of enrollment to the date of death.
Cumulative incidence of relapse (CIR) | Measured up to 1 year after the last subject has enrolled or all the subjects have finished their last EFS follow up, whichever comes first.
  CIR will be defined as the cumulative proportion of subjects who has relapsed after achieving a composite complete response (CR + CRi).

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Prof., Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No